CLINICAL TRIAL: NCT05070832
Title: Deep Hyperthermia Combined With Neoadjuvant Concurrent Radiochemotherapy for Locally Advanced Rectal Cancer, PUTHRC-001：A Multi-Center, Open-Label, Randomized Controlled Study
Brief Title: Hyperthermia Combined With Neoadjuvant Radiochemotherapy for LARC
Acronym: PUTHRC-001
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Beijing Chao Yang Hospital (Other); Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUTHRC-001
Record Dates: First submitted 2021-09-17; First posted 2021-10-07 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Hyperthermia; Radiotherapy
Keywords: locally advanced rectal cancer; hyperthermia; neoadjuvant therapy; chemoradiotherapy
MeSH Terms: conditions — Hyperthermia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperthermia Group (Experimental): The neoadjuvant therapy is hyperthermia combined with concurrent radiochemotherapy for this group.
  Interventions: Procedure: Deep Hyperthermia
- Non-hyperthermia group (No Intervention): The neoadjuvant treatment is concurrent radiochemotherapy, which is standard treatment for LARC according to the guidelines.

INTERVENTIONS:
Procedure: Deep Hyperthermia — Hyperthermia is a type of treatment in which tumor is heated to as high as 40.5-43℃ to help damage and kill cancer cells with little or no harm to normal tissue.
  Arms: Hyperthermia Group

SUMMARY:
The purpose of this study is to determine whether adding deep hyperthermia to neoadjuvant concurrent radiochemotherapy could improve T-downstaging rate for locally advanced rectal cancer (LARC).

DETAILED DESCRIPTION:
The purpose of this study is to determine whether adding deep hyperthermia to neoadjuvant concurrent radiochemotherapy could improve T-downstaging rate for locally advanced rectal cancer (LARC). The sample size is 142. Patients with LARC (T3-4/N+) will be randomly divided into intervention group and control group. For intervention group, the neoadjuvant therapy is hyperthermia combined with concurrent radiochemotherapy. For control group, the neoadjuvant treatment is concurrent radiochemotherapy. T-downstaging rate will be used to evaluate the effectiveness of deep hyperthermia. T-downstaging is defined as the postoperative pathological T stage lower than the original T stage by imaging before treatment.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Pathologically diagnosed as rectal adenocarcinoma
* Locally advanced rectal cancer (T3-4/N+) staging by CT, MRI and/or endoscopy
* Males with fertility and females of childbearing age must take effective contraceptive measures at least since signing informed consent until 180 days after the end of concurrent radiotherapy and chemotherapy. Childbearing age means pre-menopausal or within 2 years after menopause. Women of childbearing age must exclude pregnancy before concurrent radiotherapy and chemotherapy
* Patients with normal organ function prior to treatment, the following criteria are met:a) blood routine examination criteria : i) hemoglobin (HB) ≥90g/L; ii) absolute neutrophil count (ANC) ≥1.5×10e9/L; iii) platelet (PLT) ≥70×10e9/L; b) biochemical tests meet the following criteria: i) serum creatinine (Cr) ≤1.5 times of upper limit of normal (ULN) or creatinine clearance (CCr) ≥40ml/min; ii) total bilirubin (TBIL) ≤1.5 ULN; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 ULN, e）Coagulation test: International Normalized Ratio (INR)≤ 1.5 × ULN, Prothrombin Time ≤ 1.5 × ULN

Exclusion Criteria:

* Patients with signet ring cell carcinoma or mucinous adenocarcinoma.
* Patients who refuse to undergo hyperthermia or cannot cooperate with continuous follow-up.
* Patients with severe bleeding tendency, severe infection, wounds or infections on the skin of the hyperthermia area.
* Patients who have metal implants or pacemakers in their bodies who cannot tolerate excessively high temperatures.
* Other primary malignant tumors occurred within 5 years before concurrent radiotherapy and chemotherapy, except for malignant tumors that have undergone radical treatment and are locally curable (such as basal or squamous cell skin cancer, superficial bladder cancer or prostate, cervical or breast carcinoma in situ, etc.).
* Suffer from uncontrollable comorbid diseases, including but not limited to symptomatic congestive heart failure, uncontrollable hypertension, unstable angina, arrhythmia, active peptic ulcer or bleeding disease.
* Patients with a history of alcohol or drug abuse.
* Patients who do not agree to participate in this study or unable to complete the informed consent process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Tumor T-downstaging rate | 12 weeks
  T-downstaging is defined as the postoperative pathological T stage lower than the original T stage by imaging before treatment.

SECONDARY OUTCOMES:
Tumor shrinkage percentage | 12 weeks
  （tumor volume before treatment-tumor volume before neoadjuvant treatment) /（ tumor volume before neoadjuvant treatment）
Complete tumor resection rate | 12 weeks
  （patient number of R0 resection）/（total number of patients undergoing surgery）
Pathological complete response rate | 12 weeks
  （number of patients with no residual tumors after neoadjuvant therapy）/（total number of patients undergoing surgery）
Perioperative complication rate | 4 months
  （number of patients with complications before or after surgery）/（total number of patients undergoing surgery）
Anal retention rate | 12 weeks
  （number of patients with anus preservation after surgery）/（total number of patients undergoing surgery）
Disease-free survival | 3 year
  the time from random day to disease progression or death (whichever occurs first);
Overall survival | 3 year
  the time between a random day and the day of death from any cause.
36-Item Short-Form Health Survey（SF-36） | 3 year
  The minimum and maximum values of SF-36 are 30 and 150. Higher score means a better quality of life.
Quality of Life Questionnaire-Core 30（QLQ-C30） | 3year
  The minimum and maximum values of QLQ-C30 are 0 and 100. Higher score means a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Hao Wang, Doctor, Study Director — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No